CLINICAL TRIAL: NCT05841368
Title: DELIRIUM SCREENING, INCIDENCE AND MANAGEMENT OBSERVATIONAL STUDY IN 2024 - THE CZECH REPUBLIC
Acronym: DELUSION
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other); Department of Neurology, University Hospital Brno (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: DELUSION-24-CZ
Record Dates: First submitted 2023-04-22; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Delirium
Keywords: Delirium; Screening; Therapy; CAM-ICU
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult ICU patients: Adult patients in ICU setting
  Interventions: Diagnostic Test: CAM-ICU
- Pediatric ICU patients: Pediatric patients in ICU setting
  Interventions: Diagnostic Test: pCAM-ICU

INTERVENTIONS:
Diagnostic Test: CAM-ICU — Delirium in adult patients will be screened according to CAM-ICU
  Other Names: delirium screening
  Groups: Adult ICU patients
Diagnostic Test: pCAM-ICU — Delirium in adult patients will be screened according to pCAM-ICU
  Other Names: delirium screening
  Groups: Pediatric ICU patients

SUMMARY:
Delirium in intensive care unit (ICU) settings is a frequent complication with reported prevalence of 31%. Recent data has revealed the connection between delirium and increased 30days mortality after hospital release and the higher incidence of readmission to emergency. Despite the high prevalence and well described validation methods for screening, the precise incidence remains unclear due to insufficient screening in ICU settings. The incidence of delirium in Czech Republic remains undescribed, beside data reported from neurointensive care patients and single-center general critically ill patients data.

DETAILED DESCRIPTION:
All patients fulfilling inclusion criteria in intensive care settings in involved ICUs in Czech Republic will be included into the study. Data will be recorded for 1 consequent month. Basic demography will be evaluated. In each patient standard delirium screening based on the institutional ICU rules will be performed. If no screening method were set,Confusion Assessment Method - CAM-ICU for adult and pediatric Confusion Assessment Method -pCAM-ICU for pediatric patients would be used together with delirium management, restrain procedures, sedative/neuroleptics administration, 28-days mortality. All data will be recorded into to predefined eCRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU settings
* in defined time interval of the study

Exclusion Criteria:

* duration of ICU stay shorter than 24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Delirium prevalence | during 30 days after study initiation in selected ICU
  Delirium prevalence by CAM-ICU and pCAM-ICU will be screened in defined time interval

SECONDARY OUTCOMES:
Delirium management | during 30 days after study initiation in selected ICU
  Management of delirium will be evaluated
Inhospital mortality | during 30 days after study initiation in selected ICU
  Inhospital mortality will be evaluated
28-days mortality | after patient inclusion into the study
  28-days mortality will be evaluated
90-days mortality | after patient inclusion into the study
  long term mortality will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided